CLINICAL TRIAL: NCT07150273
Title: A Randomized, Single-Center, Patient & Evaluator-Blind, Matched Pairs, Active-Controlled Design Confirmatory Clinical Study to Evaluate the Efficacy and Safety of the Injection With UNIVELO Sub-Q, as Compared to Restylane® Sub-Q, in the Temporary Correction of the Nasolabial Fold
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of the Injection With UNIVELO Sub-Q, as Compared to Restylane® Sub-Q, in the Temporary Correction of the Nasolabial Fold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jetema Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO_UNI_1506
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Nasolabial Fold

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Device - UNIVELO Sub-Q (Experimental): UNIVELO Sub-Q
  Interventions: Device: UNIVELO Sub-Q 2mL
- Comparator Device - Restylane Sub-Q (Active Comparator): Restylane Sub-Q
  Interventions: Device: Restylane Sub-Q 2mL

INTERVENTIONS:
Device: UNIVELO Sub-Q 2mL — Test device
  Arms: Test Device - UNIVELO Sub-Q
Device: Restylane Sub-Q 2mL — Comparator Device
  Arms: Comparator Device - Restylane Sub-Q

SUMMARY:
A 48-week, single-center, randomized, patient & evaluator-blind, matched pairs, active-controlled, non-inferiority, confirmatory design

ELIGIBILITY:
Inclusion Criteria:

* Subjects who desire temporary improvement of both nasolabial folds and who has rated 3 or 4 on the Wrinkle Severity Rating Scale (WSRS) (the rating does not have to be the same for both sides)
* Subjects who have agreed to discontinue all dermatological treatments or procedures, including those for facial wrinkles improvement in the facial area, during the clinical trial period
* Subjects capable of understanding and complying with directions and who can participation for the full duration of the clinical trial period
* Subjects who have voluntarily decided to participate in the clinical trial and have given written consent by signing the subject informed consent form

Exclusion Criteria:

* Subjects who have been administered an antithrombotic agent (with the exception of low dosage aspirin (100mg, maximum 300mg/day)) within 2 weeks of the date of the screening
* Subjects who have had a history of any bleeding disorder, in the past or the present

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) | 24 weeks
  Measure severity of wrinkle from score of 1 (no visible fold) to 5 (extremely deep and long folds)

SECONDARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) | 8 weeks, 16 weeks, 36 weeks, 48 weeks
  Measure severity of wrinkle from score of 1 (no visible fold) to 5 (extremely deep and long folds)
Global Aesthetic Improvement Scale (GAIS) | 8 weeks, 16 weeks, 24 weeks, 36 weeks, 48 weeks
  Measure improvement status of wrinkle from score of -1 (worse) to 3 (very much improved)